CLINICAL TRIAL: NCT02713009
Title: Investigation of the Impact of Maternal Body Weight on Vitamin D Status During Pregnancy: a Randomised Supplementation Study
Brief Title: Impact of Maternal Body Weight on Vitamin D Status During Pregnancy
Acronym: MO-VITD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Western Health and Social Care Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: REC 15/NI/0068
Record Dates: First submitted 2016-01-14; First posted 2016-03-18 (Estimated); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Obesity; Vitamin D Deficiency
Keywords: Maternal body weight; Vitamin D; Pregnancy
MeSH Terms: conditions — Obesity; Vitamin D Deficiency | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment 1 (Experimental): Pregnancy multivitamin + vitamin D daily from ~Week 12 gestation until delivery
  Interventions: Dietary Supplement: Pregnancy multi-vitamin (including 10μg vitamin D3); Dietary Supplement: 10μg vitamin D3
- Treatment 2 (Placebo Comparator): Pregnancy multivitamin + placebo daily from ~Week 12 gestation until delivery
  Interventions: Dietary Supplement: Pregnancy multi-vitamin (including 10μg vitamin D3); Dietary Supplement: 0μg vitamin D (placebo)

INTERVENTIONS:
Dietary Supplement: Pregnancy multi-vitamin (including 10μg vitamin D3)
Dietary Supplement: 10μg vitamin D3
  Arms: Treatment 1
Dietary Supplement: 0μg vitamin D (placebo)
  Arms: Treatment 2

SUMMARY:
Research shows high levels of vitamin D deficiency in pregnant women in Northern Ireland. Body composition is a determinant of vitamin D status. Vitamin D is a fat soluble vitamin and therefore may be hidden within the adipose/fat tissue in overweight/obese individuals. All pregnant and breastfeeding women are advised to take a daily supplement containing 10μg vitamin D. The investigators hypothesise that overweight/ obese pregnant women have a lower vitamin D status than their leaner counterparts at the start of pregnancy and may need a higher daily supplementation to achieve a sufficient status.

The investigators propose a randomised supplementation study where pregnant women (n 240) from the Western Health and Social Care Trust Area will be invited to take part.

Inclusion criteria: pregnant women first trimester, without current pregnancy related complications, singleton pregnancy, aged ≥18 years, with Body Mass Index (BMI) > 18.5kg /m².

Participants will be randomised to receive either 0μg (placebo) plus a multivitamin or 10μg vitamin D plus a multivitamin from 12 weeks gestation until delivery. The multivitamin already contains 10μg vitamin D; Therefore participants will be randomised to receive a total of 10μg or 20μg vitamin D.

Blood samples (20mls) will be taken at 12, 28 and 36 weeks gestation. A sample of blood will be taken from the cord after delivery. Vitamin D status is the main outcome measurement. All blood samples will be analysed for vitamin D and other associated metabolites. Data will be collected on health and lifestyle, supplementation use and food intake. Body composition measurements will be recorded at each appointment and infant anthropometric measurements will be taken from the maternal notes after delivery. Findings from this research will be used to inform nutrition policy on appropriate vitamin D supplementation levels in pregnancy which may be dependent upon pre pregnancy BMI.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Age ≥18years
* BMI >18.5 kg/m²
* Without current pregnancy related complications
* At least 12 weeks gestation
* Have a singleton pregnancy (as confirmed at first scan)
* Pregnant women who are currently taking vitamin D and have had a sun holiday will be included in this study. All participants will agree to discontinue any current supplementation and will be provided with a multivitamin for the duration of pregnancy.

Exclusion Criteria:

* Aged <18 years
* Pregnancy BMI <18.5kg/m²
* Participants with multiple pregnancy
* Participants currently involved in another research study
* Participants with a history of gastrointestinal, hepatic, renal, vascular or haematological disorders.
* Participants who have had in vitro fertilisation (IVF) treatment
* Participants with a history of NTD affected pregnancies
* Pregnant women with active thyroid disease (e.g., Graves, Hashimoto or thyroiditis)
* Planned home births

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in Vitamin D (25-hydroxyvitamin D) status | Baseline (Week 12 gestation), Mid-point (Week 28 gestation) & End of pregnancy (Week 36 gestation + Delivery)
  Serum Vitamin D status (Week 12, 28 + 36 gestation) & cord serum Vitamin D status (delivery)

SECONDARY OUTCOMES:
Gestational weight gain | Baseline (Week 12 gestation), Mid-point (Week 28 gestation) & End of pregnancy (Week 36 gestation)
Change in inflammation status | Baseline (Week 12 gestation), Mid-point (Week 28 gestation) & End of pregnancy (Week 36 gestation + Delivery)
  Plasma inflammation status (Week 12, 28 + 36 gestation) & cord plasma inflammation status (delivery)
Change in bone turnover markers | Baseline (Week 12 gestation), Mid-point (Week 28 gestation) & End of pregnancy (Week 36 gestation + Delivery)
  Plasma bone turnover markers (Week 12, 28 + 36 gestation) & cord plasma bone turnover markers (delivery)
Genetics | Baseline (Week 12 gestation)
  e.g. CYP2R1, CYP27B1, CYP24A1
Dietary intake | Week 28 gestation
  Food diary with food frequency questionnaire
Foetal growth chart measurement | Baseline (Week 12 gestation), Mid-point (Week 28 gestation) & End of pregnancy (Week 36 gestation + Delivery)
Change in Vitamin D related measures | Baseline (Week 12 gestation), Mid-point (Week 28 gestation) & End of pregnancy (Week 36 gestation + Delivery)
  Blood Vitamin D related status (Week 12, 28 + 36 gestation) & cord Vitamin D related status (delivery)
Haemoglobin | Baseline (Week 12 gestation), Mid-point (Week 28 gestation) & End of pregnancy (Week 36 gestation + Delivery)
  As part of full blood count
Plasma ferritin | Baseline (Week 12 gestation), Mid-point (Week 28 gestation) & End of pregnancy (Week 36 gestation + Delivery)
  Clinical chemistry analyser
Transferrin saturation | Baseline (Week 12 gestation), Mid-point (Week 28 gestation) & End of pregnancy (Week 36 gestation + Delivery)
  Clinical chemistry analyser
Iron status | Baseline (Week 12 gestation), Mid-point (Week 28 gestation) & End of pregnancy (Week 36 gestation + Delivery)
  Serum, clinical chemistry analyser
Soluble transferrin receptor | Baseline (Week 12 gestation), Mid-point (Week 28 gestation) & End of pregnancy (Week 36 gestation + Delivery)
  ELISA
Hepcidion | Baseline (Week 12 gestation), Mid-point (Week 28 gestation) & End of pregnancy (Week 36 gestation + Delivery)
  ELISA
Methylation analysis | Baseline (Week 12 gestation), Mid-point (Week 28 gestation) & End of pregnancy (Week 36 gestation + Delivery)
  Iron and vitamin D related genes

CONTACTS AND LOCATIONS:
Locations (1):
- Western Health and Social Care Trust, Altnagelvin, Londonderry, Co.Londonderry, United Kingdom

REFERENCES:
- [Derived] Alhomaid RM, Mulhern MS, Strain J, Laird E, Healy M, Parker MJ, McCann MT. Maternal obesity and baseline vitamin D insufficiency alter the response to vitamin D supplementation: a double-blind, randomized trial in pregnant women. Am J Clin Nutr. 2021 Sep 1;114(3):1208-1218. doi: 10.1093/ajcn/nqab112. PMID 33964855